CLINICAL TRIAL: NCT04998916
Title: MPFC Theta Burst Stimulation as a Treatment Tool for Alcohol Use Disorder: Effects on Drinking and Incentive Salience
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Lisa McTeague, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00102709; 2P50AA010761-26 (NIH)
Record Dates: First submitted 2021-08-03; First posted 2021-08-10 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder; Alcohol Drinking; Substance Use; Drinking, Alcohol; Alcohol Use Disorder (AUD)
Keywords: Transcranial Magnetic Stimulation; Medial Prefrontal Cortex; Brain Stimulation; Non-invasive; Adult
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This study will utilize a double-blind, sham-controlled clinical trial to evaluate the efficacy of the TBS treatment to the vmPFC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Real TBS to the mPFC (Experimental): For continuous theta burst stimulation (cTBS), participants will receive 3 sessions of stimulation per visit over the left medial prefrontal cortex (mPFC) (each train: 3 pulse bursts presented at 5Hz, 15 pulses/sec, 600 pulses/session, 60 sec intertrain interval; 120% RMT, MagPro; 10-15 min inter session interval) using a figure 8 coil (Coil Cool-B65 A/P).
  Interventions: Device: Real TBS to the mPFC
- Sham TBS to the mPFC (Sham Comparator): The MagVenture MagPro system has an integrated, active sham which passes current through two surface electrodes placed on the scalp. The electrodes will be placed on the left frontalis muscle for all sessions. A patient identification card will randomize participants to receive either real or sham stimulation. This system maintains blinding by a gyroscope in the coil which indicates to the clinical staff whether the coil should be rotated up or down for this participant once the card is entered into the machine. One side of the coil is active, the other is sham. The integrity of the double-blind procedure will be assessed by asking the patients and study personnel rate their confidence regarding whether they thought they received real or sham (scale 1-10).
  Interventions: Device: Sham TBS to the mPFC

INTERVENTIONS:
Device: Real TBS to the mPFC — This will be delivered with the Magventure Magpro system; 600 pulses of continuous theta burst stimulation with the active sham coil (double blinded using the integrated active sham system).
  Arms: Real TBS to the mPFC
Device: Sham TBS to the mPFC — This will be delivered with the Magventure Magpro system; 600 pulses with the active sham coil (double blinded using the integrated active sham system). The MagVenture MagPro system has an integrated active sham that passes current through two surface electrodes placed on the scalp. The electrodes are placed on the left frontalis muscle under the coil for both the real and sham stimulation sessions.
  Arms: Sham TBS to the mPFC

SUMMARY:
The purpose of this study is to develop transcranial magnetic stimulation (TMS), specifically TMS at a frequency known as theta burst stimulation (TBS), to see how it affects the brain and changes the brain's response to alcohol-related pictures. TMS and TBS are stimulation techniques that use magnetic pulses to temporarily excite specific brain areas in awake people (without the need for surgery, anesthetic, or other invasive procedures). TBS, which is a form of TMS, will be applied over the medial prefrontal cortex, (MPFC), which has been shown to be involved with drinking patterns and alcohol consumption. This study will test whether TBS can be used as an alternative tool to reduce the desire to use alcohol and reducing the brain's response to alcohol-related pictures.

DETAILED DESCRIPTION:
With advances in optogenetic stimulation techniques, preclinical studies have demonstrated that activity in frontal-striatal neural circuits has a causal influence on heavy drinking and alcohol reinstatement. Clinically, however, this research has not yet been translated into a neural circuit based therapeutic technique for patients with alcohol use disorder (AUD). The long term goal of this multidisciplinary research study team is to determine the optimal parameters through which non-invasive transcranial magnetic stimulation can be used to improve alcohol drinking outcomes (abstinence, heavy drinking days) among individuals seeking behavioral treatment for AUD. Building on a foundation of several target identification studies and a small double-blinded clinical trial in treatment-engaged AUD patients performed by the study team in the Charleston Alcohol Research Center, here the investigator proposes a double-blind placebo controlled, randomized study to evaluate the efficacy of theta burst stimulation (TBS) to medial prefrontal cortex (mPFC) as a tool to decrease drinking and brain reactivity to alcohol cues among treatment-seeking individuals with AUD. Individuals will be screened initially by the Clinical Intake and Assessment core, then given an opportunity to enroll in this study, provide informed consent, and be randomized to receive real or sham TBS to the mPFC 36 sessions (3x/day on each of 3 days/week over 4 weeks, i.e., 12 days). The scientific premise of this 5 year proposal is that, by modulating the neural circuits that regulate alcohol cue-reactivity it will be possible to increase alcohol abstinence rates and decrease heavy drinking days over a 4 month period. With the combined scientific expertise in brain stimulation, neuroimaging, alcohol use disorder research in the Charleston Alcohol Research Center, and clinical practice at MUSC, the study team is uniquely suited to develop this critical line of research. The outcomes of the proposed Aims will provide an evidence-based foundation for a multisite clinical trial and will hasten progress towards developing a new neural circuit based treatment for patients with AUD.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65 (to maximize participation; note: Scalp-to-Cortex distance will be included as a covariate to calculate adjusted TMS dose given expected cortical atrophy in heavy alcohol users and older adults and the demonstrated effect50 on TMS-fMRI responses in addiction)
* Alcohol Use Disorder, determined by DSM-V criteria, using the Structured Clinical Interview for DSM-V
* Consumption of more than 14 drinks (women) or 21 drinks (men) per week, with at least 4 heavy drinking days (defined as ≥ 4 drinks for women and ≥ 5 for men) per week during the 30-days prior to enrolling.
* Able to read and understand questionnaires and informed consent.

Exclusion Criteria:

* Has metal placed above the neck
* Is at elevated risk of seizure (i.e., has a history of seizures, is currently prescribed medications known to lower seizure threshold)
* Has a history of moderate to severe alcohol withdrawal or medicated alcohol withdrawal
* Has a history of claustrophobia
* Has a history of chronic migraines
* Has a history of traumatic brain injury, including a head injury that resulted in hospitalization, loss of consciousness for more than 10 minutes, or having ever been informed that they have an epidural, subdural, or subarachnoid hemorrhage
* Has an unstable medical illness requiring planned medical/surgical intervention (e.g. chemotherapy, surgical procedure)
* Medications: Is currently taking or initiates a new prescription for drugs known to improve alcohol drinking treatment outcomes (e.g. naltrexone, acamprosate, topiramate) or taking psychiatric/sleeping medications except for stable (1 month) antidepressants/SSRI's. [Note: this criterion is for scientific rather than safety or patient comfort reasons].
* Has a history of substance use disorder (other than nicotine) by DSM-V criteria in the past 6 months
* Meets DSM V criteria for panic disorder, bipolar disorder, obsessive-compulsive disorder, schizophrenia, dissociative disorders, eating disorders, and any other psychotic disorder. [Note: The inclusion of participants with other affective and anxiety disorders is essential because of the marked frequency of the co-existence of mood and other anxiety disorders among patients with AUD at large]
* Has current suicidal ideation or homicidal ideation
* Females of childbearing potential who are pregnant (by urine HCG), nursing, or who are not using a reliable form of birth control.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Percent Heavy Drinking Days (PHDD) from baseline | Baseline (Week 1), Post-treatment (4-weeks from baseline), 1-month post treatment (Follow-up #1), 2-months post treatment (Follow-up #2), 3-months post treatment (Follow-up #3)
  The primary outcome analysis will examine the TMS treatment effect (active vs. sham) on drinking outcomes-measured as percent heavy drinking days (PHDD) (heavy drinking day defined as 4 or more drinks for women and 5 or more drinks for men)-in the follow-up period beginning after the final treatment session. Collected via timeline follow back (TLFB) in three 28-day (month) intervals, this will be analyzed using multivariate mixture models to consider the effect of time (month after treatment) and the interaction of treatment with time, baseline drinking, number of treatment sessions received, and any other potential covariates (e.g., age, nicotine use, time since last drink). Drinking data will be collected on all randomized participants, irrespective of treatment completion. Lower percentages indicate fewer heavy drinking days in the 28-day interval.
Change in Percent Days Abstinent (PDA) from baseline | Baseline (Week 1), Post-treatment (4-weeks from baseline), 1-month post treatment (Follow-up #1), 2-months post treatment (Follow-up #2), 3-months post treatment (Follow-up #3)
  The primary outcome analysis will examine the TMS treatment effect (active vs. sham) on drinking outcomes-measured as percent days abstinent (PDA) - in the follow-up period beginning after the final treatment session. Collected via timeline follow back (TLFB) in three 28-day (month) intervals, this will be analyzed using multivariate mixture models to consider the effect of time (month after treatment) and the interaction of treatment with time, baseline drinking, number of treatment sessions received, and any other potential covariates (e.g., age, nicotine use, time since last drink). Drinking data will be collected on all randomized participants, irrespective of treatment completion. Higher percentages indicate increased days abstinent from alcohol in the 28-day interval.
Change in alcohol cue task MRI activation 1-week post treatment from baseline | Baseline (Week 1), Post-treatment (4-weeks from baseline)
  For the alcohol cue reactivity task, multivariate mixture model analyses will be used to calculate the difference in activation between the ALC and BEV blocks for vmPFC and ventral striatal ROIs, and to analyze maximum likelihood estimates for ALC vs. BEV activation as a function of time, treatment, and the cross-level interactions of these factors. Specifically, the cue task stimuli will be nested within time (post- vs. pre-treatment scan); time will be nested within participant; and participants will be nested within treatment (Sham vs. Active).

SECONDARY OUTCOMES:
Change in anxiety via State-Trait Anxiety Inventory from baseline | Baseline (Week 1), Post-treatment (4-weeks from baseline), 1-month post treatment (Follow-up #1), 2-months post treatment (Follow-up #2), 3-months post treatment (Follow-up #3)
  As an exploratory analysis, anxiety will be measured using the State-Trait Anxiety Inventory to assess the impact of treatment on self-reported comorbid affective psychopathology. Scoring ranges from 20-80 for each subscale, with higher scores indicating higher anxiety symptoms.
Change in alcohol use via Obsessive-Compulsive Drinking Scale from baseline | Baseline (Week 1), Post-treatment (4-weeks from baseline), 1-month post treatment (Follow-up #1), 2-months post treatment (Follow-up #2), 3-months post treatment (Follow-up #3)
  As an exploratory analysis, alcohol craving will be measured using the Obsessive-Compulsive Drinking Scale to assess the impact of treatment on self-reported obsessive-compulsive aspects of craving. Scoring ranges from 0-40, with 0 indicating a higher ability to control drinking. This questionnaire also includes an obsessive sub-scale and a compulsive sub-scale each ranging from 0-20, with lower scores indicating lower aspects of alcohol craving and higher ability to control these urges.
Change in depression via Becks Depression Inventory-II from baseline | Baseline (Week 1), Post-treatment (4-weeks from baseline), 1-month post treatment (Follow-up #1), 2-months post treatment (Follow-up #2), 3-months post treatment (Follow-up #3)
  As an exploratory analysis, depression will be measured using the Becks Depression Inventory-II to assess the impact of treatment on self-reported comorbid affective psychopathology. Scoring ranges from 0-63, with higher scores indicating higher levels of depressive symptoms.
Change in alcohol use via Alcohol Audit from baseline | Baseline (Week 1), Post-treatment (4-weeks from baseline), 1-month post treatment (Follow-up #1), 2-months post treatment (Follow-up #2), 3-months post treatment (Follow-up #3)
  As an exploratory analysis, alcohol severity will be measured using the Alcohol AUDIT assessment to assess the impact of treatment on self-reported alcohol severity. Scoring ranges from 0-40, with 40 indicating a higher risk of alcohol severity.
Changes in cognitive performance from baseline | Baseline (Week 1), Post-treatment (4-weeks from baseline)
  Individual domains of the cognitive test battery will be tested as well as a linear composite to ascertain potential effects in specific domains as well as broader cognitive function. The same multivariate mixture model analyses will be performed on a composite measure of neurocognitive behavioral performance (assessed at baseline and end of treatment phase) to assess whether the TMS treatment affects neurocognitive performance.
Changes in Snaith-Hamilton Pleasure Scale from baseline | Baseline (Week 1), Weekly throughout treatment (Weeks 1-4), Post-treatment (4-weeks from baseline)
  The same multivariate mixture model analyses will be performed on the Snaith-Hamilton Pleasure Scale assessed weekly during treatment to examine whether hedonic tone/natural reward responsivity is influenced by active TMS.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No